CLINICAL TRIAL: NCT00173186
Title: Aortic Regurgitation After Surgical Repair of Outlet-Type Ventricular Septal Defect
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700517
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-06

CONDITIONS: Heart Septal Defects, Ventricular; Aortic Valve Insufficiency
Keywords: ventricular septal defect; aortic regurgitation
MeSH Terms: conditions — Heart Septal Defects, Ventricular; Aortic Valve Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

SUMMARY:
The major risk factors of aortic valve replacement in three outlet types VSD after surgical repair were the severity of preoperative AR and older operation age. For those patients with less than moderate degree AR preoperatively, AR progressed rarely and all in those with aortic valvar and subvalvar anomalies.

DETAILED DESCRIPTION:
Progression of aortic regurgitation (AR) in repaired outlet (juxta-arterial, muscular outlet and perimembranous outlet) ventricular septal defect (VSD) remains unclear.

From 1987 to 2002, 411 patients with complete follow-up after repair of outlet VSD constituted the study population. Study end point was aortic valve replacement or mortality.

Aortic valve replacement was performed in seventeen patients (4.1%), in whom logistic regression showed only the severity of preoperative AR and age at VSD repair as the predictors. After excluding the eleven patients with endocarditis from analysis, there were 377 patients with none to mild AR (Group I) and 23 with moderate to severe AR (Group II) preoperatively. Total follow-up was 2,230 person-years. After VSD repair, the 5- and 10-year freedom from aortic valve replacement in Group I was 100%, and in Group II 50.2%. In Group II, ten patients received aortic valve replacement and 8 underwent valvuloplasty with VSD repair. One patient needed valve replacement four years later. Age at VSD repair was the predictor for aortic valve replacement. In Group I, AR progressed in four patients (1.2%, two juxta-arterial and two perimembranous outlet) 3.5 to 7.9 years later and was associated with aortic valvar or subvalvar anomalies. The event-free curves in three outlet types VSD showed no differences.

Although AR progressed rarely (probably not in muscular outlet type) in repaired outlet types VSD with none to mild preoperative AR, in the presence of aortic valvar or subvalvar anomalies, early surgical repair of the VSD is still warranted.

ELIGIBILITY:
Inclusion Criteria:

* ventricular septal defect patients receiving total repair from Jan, 1987 to Dec, 2002.
* follow up more than 1 year after operation

Exclusion Criteria:

* complex cardiac lesions

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 411
Dates: Start 1987-01; Study Completion 2005-02

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Hwan Wu, MD, PhD, Study Chair — National Taiwan University Hospital
Locations (1):
- Department of Pediatrics, National Taiwan University Hospital, Taipei, Taiwan